CLINICAL TRIAL: NCT00240487
Title: Nitric Oxide Administration for Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-9-2088
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; ARDS; Nitric Oxide
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitric oxide first (Active Comparator): Subjects will be randomized to receive Nitric Oxide (NO) immediately after study entry, given at 10 parts per million (ppm) for the first 4 hours of study participation. Blood gases will be monitored once an hour for 4 hours. After the first 4 hours of study participation, the nitric oxide (NO) will be turned off and subjects will receive no intervention (no nitric oxide) for the next 4 hours of study participation. During this time, all subjects will receive standard clinical are. Blood gases will be monitored once an hour for 4 hours.
  Interventions: Drug: Nitric Oxide; Other: No Intervention
- Delayed nitric oxide (Active Comparator): Subjects will be randomized to receive no intervention (no nitric oxide) for he first 4 hours of study participation. During this time, all subjects will receive standard clinical care. Blood gases will be monitored once an hour for 4 hours. After the first 4 hours of study participation, the nitric oxide will be turned on and subjects will receive 10 ppm of nitric oxide for the next 4 hours of study participation. Blood gases will be monitored once an hour for 4 hours.
  Interventions: Drug: Nitric Oxide; Other: No Intervention

INTERVENTIONS:
Drug: Nitric Oxide — Subjects will receive inhaled Nitric Oxide at a dose of 10 parts per million (ppm) for a 4 hour study period. Blood gases will be collected once an hour.
  Other Names: Inhaled Nitric Oxide
Other: No Intervention — Subjects will receive no intervention (i.e., no nitric oxide treatment) for a 4 hour study period. Blood gases will be collected once an hour. During this time, all subjects will receive standard clinical care.

SUMMARY:
This research project is an open-label, randomized study for the use of Nitric Oxide in pediatric patients with acute respiratory distress syndrome (ARDS). The study examines whether nitric oxide (NO) treatment impacts the the P:F ratio (arterial partial pressure of oxygen (PaO2) divided by fraction of inspired oxygen (FiO2) in patients with ARDS. The goal of the study is to evaluate whether the order of NO therapy will have any effect on response, and evaluate the characteristics of patients who respond to NO compared to those who do not.

DETAILED DESCRIPTION:
At low concentrations, nitric oxide(NO) functions as a cellular messenger and regulator of microcirculation. NO may have an important role in the pathogenesis of ARDS as well as its treatment. NO may be primarily useful in improving matching of ventilation and perfusion in the lung. The aims of the study are to attempt to show that NO will improve oxygenation as evidenced by improvement in PaO2/FiO2. Secondary aims are to see if the improvement in oxygenation allows there to be decreased time on FiO2>0.60, evaluate whether the order of NO therapy will have any effect on response, and evaluate the characteristics of patients who respond to NO compared to those who do not.

Subjects will be randomized to receive either nitric oxide first (nitric oxide for the first 4 hours, then no intervention/no nitric oxide for the next 4 hours) or delayed treatment with nitric oxide (no intervention/no nitric oxide for the first 4 hours, then nitric oxide for the next 4 hours)..

Blood gases were monitored once an hour during study participation (total of 8 hours). Final PaO2/FiO2 levels will be compared after 8 hours of study treatment in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patient is intubated and mechanically ventilated in the Pediatric Intensive Care Unit with a PaO2/FiO2 ratio less than or equal to 100, FiO2 greater than or equal to 0.60, PEEP greater than or equal to 10, and a Murray score greater than or equal to 2.5.

Exclusion Criteria:

* Neonates (1 week to 28 days) and/or patients on extracorporeal membrane oxygenation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2000-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo I Godinez, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Pediatric Intensive Care Unit from 2000-2008.
Groups:
- Nitric Oxide First: Subjects who were randomized to receive Nitric Oxide (NO) began receiving NO immediately after study entry, given at 10 parts per million (ppm) for the first 4 hours of study participation. Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the NO was turned off and subjects received no intervention (no nitric oxide) for the next 4 hours of study participation. Blood gases were monitored once an hour for 4 hours. After the initial 8 hours of study participation, subjects remained on whichever intervention (no intervention versus 10 ppm nitric oxide) they responded best to.
- Delayed Nitric Oxide: Subjects who were randomized to receive delayed treatment with Nitric Oxide (NO) began the first 4 hours of study participation receiving no intervention (no nitric oxide). Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the NO was turned on and subjects received 10 ppm of nitric oxide for the next 4 hours of study participation. Blood gases were monitored once an hour for 4 hours.
Period: Overall Study
Arm/Group | Nitric Oxide First | Delayed Nitric Oxide
Started | 24 | 28
Completed | 24 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nitric Oxide First: Subjects received 10 ppm nitric oxide for the first 4 hours of study participation After which, the NO was turned off and subjects received no intervention (no nitric oxide) for the next 4 hours of study participation. After the initial 8 hours of study participation, subjects will remain on whichever intervention (no nitric oxide versus 10 ppm nitric oxide) they responded best to.
- Delayed Nitric Oxide: Subjects received no intervention (no nitric oxide) for the first 4 hours of study participation. After which, they received 10 ppm nitric oxide for the next 4 hours of study participation. After the initial 8 hours of study participation, subjects will remain on whichever intervention (no nitric oxide versus 10 ppm nitric oxide) they responded best to.
- Total: Total of all reporting groups
Arm/Group | Nitric Oxide First | Delayed Nitric Oxide | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 28 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.93 (6.79) | 8.06 (6.28) | 8.84 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Mean PaO2/FiO2 Ratio
Description: Arterial blood gas measurements with cooximetry to evaluate arterial partial pressure of oxygen (PaO2) and fraction of inspired oxygen (FiO2) ratio. The mean PaO2/FiO2 ratio for each group after completion 8 hour of study participation was compared
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Immediate Nitric Oxide Treatment: Subjects who were randomized to receive immediate treatment with nitric oxide (NO) began receiving NO immediately after study entry, given at 10 parts per million (ppm) for the first 4 hours of study participation. Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the nitric oxide (NO) was turned off and subjects received no intervention (no nitric oxide) for the next 4 hours of study participation. During this time, all subjects received treatment standard clinical care. Blood gases were monitored once an hour for 4 hours.
- Delayed Nitric Oxide Treatment: Subjects who were randomized to receive delayed treatment with Nitric Oxide (NO) began the first 4 hours of study participation receiving no intervention (no nitric oxide). During this time, all subjects received standard clinical care. Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the nitric oxide (NO) was turned on and subjects received 10 ppm of nitric oxide for the next 4 hours of study participation. Blood gases were monitored once an hour for 4 hours.
Arm/Group | Immediate Nitric Oxide Treatment | Delayed Nitric Oxide Treatment
Number analyzed (Participants) | 24 | 28
mmHg | 115.6 (40.6) | 115.9 (40)
Statistical Analysis 1: Comparison: Immediate Nitric Oxide Treatment vs Delayed Nitric Oxide Treatment; Differences in mean PaO2/FiO2 ratios between the two groups will help to determine whether order of therapy (immediate treatment with nitric oxide versus delayed treatment with nitric oxide) impacts outcomes; Test type: Non-Inferiority or Equivalence — The primary outcome variable is the mean PaO2/FiO2 in each group after 8 hours of study participation to determine whether timing of treatment with nitric oxide impacts outcome (immediate treatment versus delayed treatment); p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: All subjects were followed for 8 hours during study participation.
Groups:
- Immediate Treatment With Nitric Oxide: Subjects who were randomized to receive immediate treatment with nitric oxide (NO) began receiving NO immediately after study entry, given at 10 parts per million (ppm) for the first 4 hours of study participation. Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the nitric oxide (NO) was turned off and subjects received no intervention (no nitric oxide) for the next 4 hours of study participation. During this time, all subjects received standard clinical care. Blood gases were monitored once an hour for 4 hours.
- Delayed Treatment With Nitric Oxide: Subjects who were randomized to receive delayed treatment with Nitric Oxide (NO) began the first 4 hours of study participation receiving no intervention (no nitric oxide). During this time, all subjects received standard clinical care. Blood gases were monitored once an hour for 4 hours. After the first four hours of study participation, the NO was turned on and subjects received 10 ppm of nitric oxide for the next 4 hours of study participation. Blood gases were monitored once an hour for 4 hours.
Arm/Group | Immediate Treatment With Nitric Oxide | Delayed Treatment With Nitric Oxide
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

LIMITATIONS AND CAVEATS:
There may be some confounding of effects of lung recruitment from high mean airway pressures over the duration of the observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No